CLINICAL TRIAL: NCT03567655
Title: Phase II Study of Fertility-sparing Management Using High-dose Oral Progestin in Young Women With Stage I Endometrial Adenocarcinoma With Grade 2 Differentiation or Superficial Myomectomy Invasion
Brief Title: Fertility-sparing Management Using High-dose Oral Progestin in Young Women With Endometrial Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Asan Medical Center (Other)
Collaborators: Korean Gynecologic Oncology Group (Other)
Responsible Party: Principal Investigator, Jeong-Yeol Park, Clinical associate professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KGOG 2020
Record Dates: First submitted 2018-04-03; First posted 2018-06-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Endometrial Cancer
Keywords: medroxyprogestrone acetate
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Medroxyprogesterone Acetate

STUDY DESIGN:
Intervention Model Description: This study is a single arm, prospective multi-institutional study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single group (Experimental): Farlutal tab. 500mg/ Pfizer to be administered
  Interventions: Drug: Farlutal tab. 500mg/ Pfizer

INTERVENTIONS:
Drug: Farlutal tab. 500mg/ Pfizer — Medroxyprogesterone Acetate

SUMMARY:
This registry aims to evaluate the efficacy of using high-dose oral progestin in young women with stage I endometrial adenocarcinoma with grade 2 differentiation or superficial myometrial invasion as a fertility-sparing management.

DETAILED DESCRIPTION:
The standard treatment for endometrial cancer is total hysterectomy and bilateral salpingo-oophorectomy, peritoneal cytology, and lymph node dissection. However, young patients who desire to preserve their potential for fertility may find this standard treatment difficult to accept. Therefore, the conservative treatment for these patients has remained a challenge. A number of studies have reported the effectiveness of hormonal therapy using systemic progestin in women clinically diagnosed with early endometrial adenocarcinoma at stage IA, grade 1, who want to maintain reproductive potential. However, there have been few prospective studies about hormonal therapy in young women with stage I endometrial adenocarcinoma with grade 2 differentiation or superficial myometrial invasion as a fertility-sparing management.

[Primary endpoint]: To evaluate the complete response rate [Sencondary endpoint]: To evaluate of disease-free survival rate, fertility outcomes and side effects of high-dose oral progestin.

To analyze predictive and prognostic biomarkers and clinicopathologic factors about response and recurrence after therapy, To analyze patient-reported outcomes.

[TREATMENT METHODS] Patients with histologically confirmed grade 1 endometrioid adenocarcinoma with superficial myometrial invasion or patients with histologically confirmed grade 2 endometrioid adenocarcinoma that is presumably confined to the endometrium or patients with histologically confirmed grade 2 endometrioid adenocarcinoma with superficial myometrial invasion are administered medroxyprogesterone Acetate(MPA) at a dosage of 500 mg/day for 12 months.

Follow-up and treatment response assessment were implemented at a 3-month interval with MRI and dilatation and curettage (D&C) procedure. The biopsy findings are compared.

[INVESTIGATIONAL PRODUCT] General Name/Brand name:Farlutal tab. 500mg/ Pfizer

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed grade 1 endometrioid adenocarcinoma with superficial myometrial invasion based on Magnetic resonance image(MRI)
* Patients with histologically confirmed grade 2 endometrioid adenocarcinoma that is presumably confined to the endometrium based on MRI
* Patients with histologically confirmed grade 2 endometrioid adenocarcinoma with superficial myometrial invasion based on MRI
* Patients who desire to preserve fertility potential
* Patients signed the written informed consent voluntarily

Exclusion Criteria:

* Patients who have severe underlying disease or complication
* Under treatment of metastatic cancer from other organs or less than 5 years after previous cancer therapy
* Acute liver disease or kidney disease
* Thrombosis or phlebothrombosis requiring treatment, Hyperlipidemia, Smoker

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Estimated)
Dates: Start 2018-07-15 (Estimated); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
complete response rate | 12 months of taking oral MPA
  Patients with histologically confirmed grade 1 endometrioid adenocarcinoma with superficial myometrial invasion or patients with histologically confirmed grade 2 endometrioid adenocarcinoma that is presumably confined to the endometrium or patients with histologically confirmed grade 2 endometrioid adenocarcinoma with superficial myometrial invasion are administered medroxyprogesterone Acetate(MPA) at a dosage of 500 mg/day for 12 months.

SECONDARY OUTCOMES:
disease-free survival | every 3 months during 24 months from time of obtaining complete response
  After obtaining complete response, this study aims to evaluate disease-free survival. The disease-free survival (DFS) time is defined as the time from the date of cancer diagnosis to the date of recurrence or date of the last known follow-up investigation.
fertility outcomes | every 3 months during 24 months from time of obtaining complete response
  After obtaining complete response, this study aims to evaluate fertility outcomes. Fertility outcomes include menstruation history ( interval , duration , amount ), pregnancy try (date/ with or without assisted reproductive technology ), the number of pregnancy and the number of live birth.
Side effects of MPA, dosage of 50mg/day | From date of starting of MPA until the study end assessed up to 36 months
  this study aims to evaluate the side effects of MPA, dosage of 50mg/day with treatment-related adverse events as assessed by CTCAE version4.0

CONTACTS AND LOCATIONS:
Overall Officials: Yong-Man Kim, MD Ph.D., Study Chair — Korean Gynecologic Oncologic Group
Locations (1):
- Department of Obstetrics and Gynecology, University of Ulsan College of Medicine, Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park JY, Nam JH. Progestins in the fertility-sparing treatment and retreatment of patients with primary and recurrent endometrial cancer. Oncologist. 2015 Mar;20(3):270-8. doi: 10.1634/theoncologist.2013-0445. Epub 2015 Feb 11. PMID 25673106
- [Background] Bokhman JV, Chepick OF, Volkova AT, Vishnevsky AS. Can primary endometrial carcinoma stage I be cured without surgery and radiation therapy? Gynecol Oncol. 1985 Feb;20(2):139-55. doi: 10.1016/0090-8258(85)90135-0. PMID 3972284
- [Background] Kempson RL, Pokorny GE. Adenocarcinoma of the endometrium in women aged forty and younger. Cancer. 1968 Apr;21(4):650-62. doi: 10.1002/1097-0142(196804)21:43.0.co;2-p. No abstract available. PMID 5643760
- [Background] Skouby SO. The rationale for a wider range of progestogens. Climacteric. 2000 Dec;3 Suppl 2:14-20. PMID 11379382